CLINICAL TRIAL: NCT04942834
Title: Using Cryoballoon Ablation as Initial Treatment for Patients With Persistent Atrial Fibrillation Comparing to Anti-arrhythmic Drugs
Brief Title: Using Cryoballoon Ablation as Initial Treatment for Persistent Atrial Fibrillation
Acronym: Cryo-InitialAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cryo-initial-AF
Record Dates: First submitted 2021-06-17; First posted 2021-06-29 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2023-08

CONDITIONS: Atrial Fibrillation, Persistent; Arrhythmias, Cardiac
Keywords: cryoablation; pulmonary vein isolation; atrial fibrillation; Anti-Arrhythmic Agents
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Sotalol; Dronedarone; Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug treatment group (Active Comparator): receive class I or class III AAD to restore or maintain sinus rhythm.
  Interventions: Drug: Antiarrhythmic drug including Propafenone, Sotalol, Dronedarone and Amiodarone
- cryoballoon ablation group (Experimental): receive cryoballoon ablation to restore sinus rhythm.
  Interventions: Device: cryoballoon ablation

INTERVENTIONS:
Drug: Antiarrhythmic drug including Propafenone, Sotalol, Dronedarone and Amiodarone — Class I or III antiarrhythmic drug, including sotalol
  Arms: Drug treatment group
Device: cryoballoon ablation — Pulmonary vein isolation by cryoballoon ablation using Medtronic Arctic Front Advance™ Cardiac CryoAblation Catheters (23mm and 28mm)
  Arms: cryoballoon ablation group

SUMMARY:
This study is to assess the effectiveness and safety of using cryoballoon ablation comparing with anti-arrhythmic drug therapy as initial treatment for naive patients with persistent atrial fibrillation.

DETAILED DESCRIPTION:
Subjects with persistent atrial fibrillation with no history of treatment with anti-arrhythmic drugs are randomized 1:1 to either an anti-arrhythmic drug or pulmonary vein isolation using the cryoballoon catheter.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of symptomatic persistent AF: Defined as having a continuous episode lasting longer than 7 days but less than 1 year documented by consecutive ECG recordings OR Defined as having a continuous episode lasting longer than 7 days but less than 1 year documented by an ECG recording and one doctor note indicating patient had symptoms consistent with AF
* Age 18 -75 years old
* Structurally normal heart with LVEF ≥50%, interventricular septum thickness ≤ 12 mm, and left atrial diameter <46 mm (short axis) as obtained by transthoracic echocardiography. •
* Normal ECG parameters when measured in sinus rhythm (QRS width ≤120 ms in a 12-channel surface ECG, QTc interval <440 ms, and PQ interval ≤210 ms).

Exclusion Criteria:

* History of AF treatment with class I or III antiarrhythmic drug, including sotalol, with the intention to prevent an AF recurrence. However, patients pretreated with above AAD for less than 7 days with the intention to convert an AF episode are allowed.
* left atrial ablation or surgical procedure (including left atrial appendage closures)
* Presence or likely implant of a permanent pacemaker, biventricular pacemaker, loop recorder, or any type of implantable cardiac defibrillator (with or without biventricular pacing function) within 12 months
* Presence of any pulmonary vein stents
* Presence of any pre-existing pulmonary vein stenosis
* Pre-existing hemidiaphragmatic paralysis
* Presence of any cardiac valve prosthesis
* +3 and +4 mitral valve regurgitation or stenosis
* Any cardiac surgery, myocardial infarction, percutaneous coronary intervention (PCI) / percutaneous transluminal coronary angioplasty (PTCA) or coronary artery stenting which occurred during the 3 month interval preceding e consent date
* Unstable angina
* New York Heart Association (NYHA) Class II, III or IV congestive heart failure
* Primary pulmonary hypertension
* Rheumatic heart disease
* Thrombocytosis, thrombocytopenia
* Any condition contraindicating chronic anticoagulation
* Active systemic infection
* Hypertrophic cardiomyopathy
* Cryoglobulinemia
* Uncontrolled hyperthyroidism
* Any cerebral ischemic event (strokes or transient ischemic attacks (TIAs)) which occurred during the 6 month interval preceding the consent date
* Any woman known to be pregnant or breastfeeding.
* Life expectancy less than one year
* Current or anticipated participation in any other clinical trial of a drug, device or biologic during the duration of the study not pre-approved by Medtronic
* Active intracardiac thrombus
* Known drug or alcohol dependency
* Unwilling or unable to comply fully with study procedures and follow-up
* Significant Chronic Kidney Disease-estimated Glomerular Filtration Rate(CKD-eGFR) <30umol/L

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Treatment success at 12 months | Randomization to 12 months
  Treatment success at 12 months after antiarrhythmic drug (AAD) initiation or ablation utilizing cryoballoon catheter measured by freedom from AF recurrence following a 3-month period after the index ablation or AAD initiation.
Rate of serious adverse events | Randomization to 12 months
  Rate of serious procedure-related and serious cryoablation system-related reported adverse events through 12 months after the index ablation procedure

SECONDARY OUTCOMES:
Quality of life changes at 12 months measured by AFEQT | one year
  The improvement in quality of life between baseline and 12 months after the index ablation procedure or AAD measured by AF Quality of Life Survey (AFEQT)
Quality of life changes at 12 months measured by SF-12 | one year
  The improvement in quality of life between baseline and 12 months after the index ablation procedure or AAD measured by 12-Item Short Form Survey (SF-12)
Arrhythmia recurrence during blanking period | 3 months
  atrial tachycardia recurrence rate during the blanking period
time to first time cardiovascular hospitalization (month) | one year
  time to first time cardiovascular hospitalization after treatment (month)

CONTACTS AND LOCATIONS:
Overall Officials: Li-qun Wu, MD,PhD, Principal Investigator — Ruijin Hospital
Locations (17):
- China (17):
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - The Affiliated Hospital Of Guizhou Medical University, Guiyang, Guizhou
  - Nanjing Drum Tower hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Affiliated Hospital Of Nantong University, Nantong, Jiangsu
  - Jiangsu Taizhou People's Hospital, Taizhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Qilu Hospital Of Shandong University, Jinan, Shangdong
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - "West China School of Medicine /West China Hospital of Sichuan University ", Chengdu, Sichuan
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - The Second Hospital Of Tianjin Medical University, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No